CLINICAL TRIAL: NCT01506843
Title: Clinical Efficacy and Mucosal/Systemic Antibody Response Changes After Sublingual Immunotherapy in Mite-allergic Children in a Randomized Double-blind, Placebo-controlled Study in Brazil
Brief Title: Sublingual Immunotherapy in Children With Allergic Rhinitis
Acronym: SLIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Ernesto Akio Taketomi, Principal Investigator, Federal University of Uberlandia
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F3046; CNPq (Other Grant/Funding Number: CNPq480010/2007-2)
Record Dates: First submitted 2011-12-20; First posted 2012-01-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2007-08

CONDITIONS: Allergic Rhinitis
Keywords: IgA antibody; IgE antibody; IgG1/IgG4 subclasses; Mite allergy; Sublingual immunotherapy; Saliva
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- mite allergen drop (Active Comparator): Children with allergic rhinitis sensitized with dust mites will receive progressive doses of allergen drops comparing those receiving placebo.
  Interventions: Biological: Mite, Mite and Bacterial or Placebo
- mite plus bacterial extracts (Active Comparator): Vaccine constituted with mite and bacterial extracts will be compared to placebo.
  Interventions: Biological: Mite, Mite and Bacterial or Placebo
- Placebo (Placebo Comparator): Placebo will be constituted by the same solution used to make dilution of the allergen extracts.
  Interventions: Biological: Mite, Mite and Bacterial or Placebo

INTERVENTIONS:
Biological: Mite, Mite and Bacterial or Placebo — All treatments were given by sublingual route according to schedule of EAACI, with some modification. Patients received up-dosing sublingual drops once a day, reaching in approximately 3 months a monthly maintenance dose of 36 μg of Der p 1 given three times a week in alternate days for mite, mite and bacterial allergen extract, and no Der p 1 and no bacterial components in the placebo group. Doses were delivered by using vials equipped with a metered-dose dropper, and subjects were instructed to hold the solution under the tongue for 2 min and not to eat or drink for 60 min after the dose. Subjects self-administered the treatment at home. Adjustments in the schedule were made on an individual basis according to standard guidelines for specific immunotherapy
  Other Names: mite allergen extract; bacterial allergen extract

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and mucosal/systemic antibody response changes after SLIT using house dust mite allergen with or without bacterial extracts in mite-allergic children.

DETAILED DESCRIPTION:
Patients with allergic rhinitis with or without asthma were selected for a randomized double-blind, placebo-controlled trial and distributed into three groups: DPT (Dpt allergen extract, n=34), DPT+MRB (Dpt allergen plus mixed respiratory bacterial extracts, n=36), and Placebo (n=32). Clinical evaluation and immunological analyses are being carried out before and after 12 and 18 months of treatment, including rhinitis/asthma symptom and medication scores, skin prick test (SPT) to Dpt, and measurements of Dpt-, Der p 1-, Der p 2-specific serum IgE, IgG4, IgG1 and -specific salivary IgA.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of allergic rhinitis
* Positive skin test to Dermatophagoides pteronyssinus total extract
* Positive serum levels of specific IgE to D. pteronyssinus extract

Exclusion Criteria:

* Previous allergen immunotherapy
* Use of antihistamines 1 week or topical corticosteroid up to 3 weeks prior to skin prick test
* Long term use of systemic corticosteroid.
* Airway infection 30 days prior to the selection.
* Children with severe asthma, malignant, cardiovascular or autoimmune diseases, under chemotherapy or immunosuppressor therapy.
* Users of cigarette smoke
* Presence of severe skin lesions

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Symptom and Medication Scores at 12 months | Baseline and 12 months
  For clinical evaluation will be used a questionnaire determining the symptom and medication scores.

SECONDARY OUTCOMES:
Change from Baseline in Specific Antibody Levels. | Baseline, 12 months and 18 Months
  Measurement of serum specific antibodies (IgE, IgG1, IgG4, and IgA) to Dermatophagoides pteronyssinus total extract, and Der p 1 and Der p 2 allergens.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto A Taketomi, MD, PhD, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Asthma and Rhinitis Control Program, Itumbiara, Goiás, Brazil